CLINICAL TRIAL: NCT06564805
Title: Clinical Trial on the Efficacy of Intralesional Triamcinolone Versus Candida Albicans Antigen in Treating Alopecia Areata
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Erika Lizbeth Alba Rojas, Erika Alba Rojas, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DE24-00008
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intralesional Triamcinolone (Active Comparator): Triamcinolone acetonide will be administered intralesionally at a concentration of 4 mg/mL. The solution will be injected in 0.1 mL doses, spaced 1 cm apart. The maximum total dose per session will be limited to 3 mL
  Interventions: Drug: Candida Albicans Antigen Injection
- Candida albicans antigen (Experimental): Single subcutaneous administration of 0.1 mL of Candida albicans antigen into one of the alopecic patches
  Interventions: Drug: Candida Albicans Antigen Injection

INTERVENTIONS:
Drug: Candida Albicans Antigen Injection — subcutaneous administration of Candida albicans antigen

SUMMARY:
The efficacy of two intralesional treatment modalities for alopecia areata will be determined. Thirty patients over the age of 6 with the diagnosis of alopecia areata on the scalp, with an extension of less than 50%, will be included. A comparison will be made between the effectiveness of intralesional Triamcinolone (standard first-line treatment) and intralesional Candida albicans antigen, with serial clinical and trichoscopic pictures at follow-up to evaluate the clinical response and associated adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alopecia areata
* SALT score of less than 50% extension
* Has not received any topical or systemic treatment in the last month
* Signed informed consent

Exclusion Criteria:

* Any skin condition on the scalp (infectious, inflammatory or neoplastic) that could modify the clinical of trichoscopic features
* Pregnancy or breast-feeding
* Patients in medications that could cause hair loss as side-effects

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment response | 5 months
  porcentage of hair growth determined by SALT score

SECONDARY OUTCOMES:
Side effects | 5 months
  Side effects associated to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fania Muñoz Garza, PhD, Principal Investigator — Hospital Universitario "Dr. José E. González"
Locations (1):
- Hospital Universitario "Dr. José Eleuterio González", Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The database with the main clinical and trichoscopic results could be shared